CLINICAL TRIAL: NCT05169593
Title: Prevention of Postoperative Endoscopic Recurrence with Endoscopy-driven Versus Systematic Biological Therapy: a Randomized, Multicentre, Parallel Group Pragmatic Non-inferiority Trial in Crohn Disease
Brief Title: Prevention of Postoperative Endoscopic Recurrence with Endoscopy-driven Versus Systematic Biological Therapy
Acronym: SOPRANO-CD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: s62015
Record Dates: First submitted 2021-11-08; First posted 2021-12-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Crohn Disease
Keywords: biological therapy; ileocolonoscopy; ileocolonic resection; ileocolonic anastomosis
MeSH Terms: conditions — Crohn Disease | interventions — Biological Products; risankizumab; vedolizumab; Ustekinumab; Infliximab; Adalimumab

STUDY DESIGN:
Intervention Model Description: A randomized, multicentre, parallel group pragmatic non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopy-driven postoperative biological therapy (Other): Endoscopic recurrence at week 30
  Adalimumab: 160 mg SC at week 32, 80 mg SC at week 34, 40 mg SC at week 36 and every two weeks thereafter.
  Infliximab: Induction with 5 mg/kg IV at week 32, and 5 mg/kg IV at week 34; maintenance with 5 mg/kg IV at week 38, week 42 or week 46 and every eight weeks thereafter or with 120 mg SC at week 38 and every two weeks thereafter.
  Ustekinumab: 260 mg (body weight ≤55kg) or 390 mg (55-85kg) or 520 mg (>85kg) IV at week 32, 90 mg SC at week 40, and every eight weeks thereafter.
  Vedolizumab: Induction with 300 mg IV at week 32, and 300 mg IV at week 34; maintenance with 300 mg IV at week 38 and every eight weeks thereafter or with 108 mg SC at week 38, week 42 or week 46 and every two weeks thereafter.
  Risankizumab: Induction with 600 mg IV at week 32, week 36 and week 40; maintenance with 360 mg SC at week 44 and every eight weeks thereafter.
  Interventions: Drug: Biological Drug
- Systematic postoperative prophylaxis with a biological (Active Comparator): Adalimumab: 160 mg subcutaneous (SC) at day 0, 80 mg SC at week 2, 40 mg SC at week 4 and every two weeks thereafter.
  Infliximab: Induction with 5 mg/kg intravenous (IV) at day 0, and 5 mg/kg IV at week 2; maintenance with 5 mg/kg IV at week 6, week 10 or week 14 and every eight weeks thereafter or with 120 mg SC at week 6 and every two weeks thereafter.
  Ustekinumab: 260 mg (body weight ≤55kg), 390 mg (55-85kg) or 520 mg (>85kg) IV at day 0, 90 mg SC at week 8 and every eight weeks thereafter.
  Vedolizumab: Induction with 300 mg IV at day 0, and 300 mg IV at week 2; maintenance with 300 mg IV at week 6 and every eight weeks thereafter or with 108 mg SC at week 6, week 10 or week 14 and every two weeks thereafter.
  Risankizumab: Induction with 600 mg IV at day 0, week 4 and week 8; maintenance with 360 mg SC at week 12 and every eight weeks thereafter.
  Interventions: Drug: Biological Drug

INTERVENTIONS:
Drug: Biological Drug — Biological therapy used in daily clinical practice in patients with Crohn's disease to prevent disease recurrence
  Other Names: Risankizumab; Vedolizumab; Ustekinumab; Infliximab; Adalimumab

SUMMARY:
With this prospective, randomized, multicentre, parallel group pragmatic non-inferiority trial, the investigators will evaluate if endoscopy-driven introduction of biological therapy is not leading to more postoperative endoscopic recurrence at week 86 compared to systematic prophylactic biological therapy in patients with CD undergoing an ileocolonic resection with ileocolonic anastomosis. Secondary analyses will include influence on clinical, biological and surgical CD recurrence, serious adverse events, direct costs, work productivity, and quality of life. If the investigators can demonstrate the non-inferiority of an endoscopy-driven approach, this patient-tailored management could be advocated, while a more expensive systematic introduction of biological therapies could be limited.

Finally, endoscopic images provided through the SOPRANO CD study, will be used to develop a new scoring system evaluating postoperative endoscopic recurrence.

DETAILED DESCRIPTION:
This will be a prospective, randomized, parallel group, pragmatic trial.

Prior to study group assignment, the type of biological therapy to be (eventually) used in the postoperative phase will be selected by the treating physician after thorough discussion with the patient. The use of cheaper anti-TNF biosimilars will be encouraged, but patients who received adalimumab and/or infliximab preoperatively cannot receive the same treatment again in SOPRANO CD if the participants previously encountered immunogenicity issues to this treatment.

Systematic postoperative prophylaxis with a biological:

Biological therapy (adalimumab, infliximab, ustekinumab, vedolizumab or risankizumab) will be initiated within 14 to 40 days after ileocolonic resection or restoration of the faecal stream (day 0).

In patients with both Harvey-Bradshaw Index (HBI) based clinical recurrence (HBI >4) and endoscopic recurrence (Rutgeerts score ≥i2b) at week 30, biological therapy will be optimized (reimbursed or through the available free goods / samples programs).

Beyond week 32 optimization of this biological therapy will be allowed following daily clinical practice including proactive therapeutic drug monitoring. However, the timing, type and reason for dose optimization should be recorded.

Endoscopy-driven postoperative biological therapy:

No CD related therapy will be administered between Baseline (14 to 40 days after ileocolonic resection or restoration of the faecal stream) and the endoscopic evaluation at week 30 Patients with endoscopic recurrence (Rutgeerts score ≥i2b) at week 30 will initiate biological therapy (adalimumab, infliximab, ustekinumab, vedolizumab or risankizumab) following a classical induction and maintenance schedule. The type of biological therapy has to be decided already in the perioperative phase to allow a proper stratification.

In patients initiating biological therapy at week 30, this therapy maybe optimized from week 32 onwards following daily clinical practice including proactive therapeutic drug monitoring. However, the timing, type and reason for dose optimization should be recorded.

In patients not on biological therapy yet but developing clinical recurrence (HBI >4) with objective signs of disease recurrence (faecal calprotectin >250 µg/g, C-reactive protein >5 mg/L or endoscopic recurrence ≥i2b or clear radiological disease activity at the neo-terminal ileum) beyond week 32, biological therapy can be initiated, but this will be regarded as a study failure.

Randomization:

Eligible patients will be allocated to one of the two treatment arms (1:1) according to a computer generated randomisation list in REDCap.

Stratified randomisation will be performed to achieve approximate balance for:

* Type of selected postoperative prophylactic therapy: adalimumab, infliximab, ustekinumab, vedolizumab or risankizumab.
* Number of risk factors for postoperative recurrence: 1, 2 or >2 (out of 5 predefined factors: active smoking, penetrating disease, previous ileocolonic resection ≤10 years of index surgery, ≥2 previous ileocolonic resections, biological therapy ≤3 months of index ileocolonic resection)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures.
2. Patients with a diagnosis of Crohn's disease based on radiology, endoscopy and/or histology
3. Males and females 18-80 years old.
4. Patients undergoing an ileocolonic resection with ileocolonic anastomosis (with or without temporary ileostomy) within 3 and 40 days prior to the Screening visit.

   Patients who underwent an ileocolonic resection with ileocolonic anastomosis with a temporary ileostomy are also eligible if the ileocolonic resection was performed within eight months prior to the Screening visit, and the restoration of the faecal stream was performed within 3 and 40 days prior to the Screening visit.
5. Patients having an increased risk for postoperative recurrence for any of the following reasons:

   1. Penetrating disease as reason for ileocolonic resection
   2. Previous ileocolonic resection within ten years of index surgery
   3. Two or more previous ileocolonic resections
   4. Active smoking
   5. Biological therapy for Crohn's disease within 3 months of index ileocolonic resection
6. Curative ileocolonic resection. All inflamed colon segments should have been removed. Strictureplasties in the small bowel not involving the anastomotic region are allowed.
7. Patients previously failing at least three months of steroids and/or three months of immunosuppressive therapy, or showing intolerance or a real contraindication for any of these therapies.
8. Patients able and willing to start and continue biological therapy, and this at the timepoint indicated through study randomization

Exclusion Criteria:

1. Participant has a history of primary non response or secondary loss of response to all five biological therapies of interest, namely adalimumab, infliximab, ustekinumab, vedolizumab and risankizumab..
2. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
3. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial.
4. Participation in an interventional Trial with an Investigational Medicinal Product (IMP) or device.
5. Patients initiating biological therapy for CD as part of another clinical trial or a medical need program.
6. Patients not understanding Dutch, French, German or English.
7. Patients with ulcerative colitis or inflammatory bowel disease type unclassified.
8. Patients with an ileorectal anastomosis, or an ileal pouch-anal anastomosis.
9. Patients with active perianal disease.
10. Patients with a colorectal stenosis.
11. Patients with an ostomy.
12. Patients with sepsis or other postoperative complications necessitating the use of antibiotics for more than ten days after ileocolonic resection or restoration of the faecal stream.
13. Patients with (an imminent risk) of a short bowel syndrome.
14. Patients who had qualifying ileocolonic resection for dysplasia or cancer without ongoing inflammation.
15. Patients with liver test abnormalities (aspartate transaminase, alanine transaminase, alkaline phosphatases, or bilirubin > 2 upper limit of normal), leukopenia (<3000 white blood cells 109/L, <1500 neutrophils 109/L ), thrombocytopenia (platelets < 50.000/mm3).
16. Patients with severe renal, pulmonary or cardiac disease.
17. Ongoing alcohol or substance abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
postoperative endoscopic recurrence (Rutgeerts score ≥i2b) | 86 weeks
  To compare the postoperative endoscopic recurrence rate in patients with Crohn's disease undergoing an ileocolonic resection with ileocolonic anastomosis randomized to systematic biological therapy or endoscopy-driven biological therapy
need for unscheduled treatment adaptation prior to week 86 | 86 weeks
  When, due to clinical symptoms, therapy needs to be started or switched prior to week 86

SECONDARY OUTCOMES:
Harvey Bradshaw Index (HBI) based clinical recurrence | 86 weeks
  HBI based clinical recurrence (score higher than 4) prior to week 86. HBI based clinical recurrence is defined as HBI >4; AND objective signs of disease recurrence, namely faecal calprotectin >250 µg/g, CRP >5 mg/L, or endoscopic recurrence Rutgeerts score ≥i2b, or clear radiological disease activity at the neo-terminal ileum.
Direct costs | 86 weeks
  Direct costs from Baseline to week 86
new ileocolonic resection | 86 weeks
  Need for a new ileocolonic resection prior to week 86
Severe adverse reactions | 86 weeks
  Severe adverse reactions to biological therapy prior to week 86
Serious adverse events | 86 weeks
  Serious adverse events prior to week 86
European Quality of Live Five Dimension Five Level Scale | 86 weeks
  Quality of life at week 30, week 62 and week 86 in comparison to Baseline (score between 0 and 100; higher score, better quality of life)

OTHER OUTCOMES:
Crohn's disease activity index (CDAI) based clinical recurrence | 86 weeks
  CDAI based clinical recurrence prior and at week 86 and time to CDAI based clinical recurrence
Harvey Bradshaw Index (HBI score higher than 4) based clinical recurrence | 86 weeks
  HBI based clinical recurrence at week 86 and time to HBI based clinical recurrence. HBI based clinical recurrence is defined as HBI >4; AND objective signs of disease recurrence, namely faecal calprotectin >250 µg/g, CRP >5 mg/L, or endoscopic recurrence ≥i2b, or clear radiological disease activity at the neo-terminal ileum.
Two-component Patient Reported Outcome (PRO-2) based clinical recurrence | 86 weeks
  PRO-2 based clinical recurrence prior and at week 86 and time to PRO-2 clinical recurrence. PRO-2 based clinical recurrence is defined as average liquid or very soft stool frequency of >2.8 and/or abdominal pain score >1.0
Endoscopic disease activity | 86 weeks
  Endoscopic disease activity (Rutgeerts score ≥i3, ≥i2a, or ≥i1) at week 86
Endoscopic recurrence | 30 weeks
  Endoscopic recurrence (Rutgeerts score ≥i2b) at week 30
Endoscopic disease activity | 30 weeks
  Endoscopic disease activity (Rutgeerts score ≥i3, ≥i2a, or ≥i1) at week 30
Persistent endoscopic recurrence | 86 weeks
  Persistent endoscopic recurrence at week 86 after development of endoscopic recurrence at week 30
a new ileocolonic resection, a balloon dilation or a strictureplasty | 86 weeks
  Need for a new ileocolonic resection, a balloon dilation or a strictureplasty at the site of the ileocolonic anastomosis prior to week 86
Work Productivity and Activity Impairment in Crohn's Disease questionnaire | 86 weeks
  Work productivity and activity impairment at week 30, week 62 and week 86 in comparison to Baseline (score between 0 and 20; lower score, better outcome)
Change in medical therapy | 86 weeks
  Change in medical therapy for Crohn's disease prior to week 86
Change in C-reactive protein | 86 weeks
  Change CRP at week 14, week 30, week 46, week 62 and week 86 in comparison to baseline
Change in faecal calprotectin | 86 weeks
  Change in faecal calprotectin at week 14, week 30, week 46, week 62 and week 86 in comparison to baseline
unscheduled visits | 86 weeks
  Number of unscheduled visits related to CD (clinical visit, endoscopic or radiological evaluation)
Suspected unexpected serious adverse reactions | 86 weeks
  Suspected unexpected serious adverse reactions prior to week 86
Two-component Patient Reported Outcome (PRO-2) based clinical recurrence in longterm follow-up | 242 weeks
  Evolution of PRO-2 at week 138, 190 and 242 in comparison to Baseline and Week 86
European Quality of Live Five Dimension Five Level Scale in longterm follow-up | 242 weeks
  Evolution of EQ-5D 5L at week 138, 190 and 242 in comparison to Baseline and Week 86
Work Productivity and Activity Impairment in Crohn's Disease questionnaire in longterm follow-up | 242 weeks
  Evolution of WPAI:CD at week 138, 190 and 242 in comparison to Baseline and Week 86
Change in C-reactive protein in longterm follow-up | 242 weeks
  Evolution of CRP at week 138, 190 and 242 in comparison to Baseline and Week 86
Change in faecal calprotectin in longterm follow-up | 242 weeks
  Evolution of faecal calprotectin at week 138, 190 and 242 in comparison to Baseline and Week 86
Change in medical therapy in longterm follow-up | 242 weeks
  Change in medical therapy for Crohn's disease prior to week 138, 190 and 242
a new ileocolonic resection, a balloon dilation or a strictureplasty in longterm follow-up | 242 weeks
  Need for a new ileocolonic resection, a balloon dilation or a strictureplasty at the site of the ileocolonic anastomosis prior to week 138, 190 and 242
Severe adverse reactions in longterm follow-up | 242 weeks
  Severe adverse reactions to biological therapy prior to week 138, 190 and 242
Serious adverse events in longterm follow-up | 242 weeks
  Serious adverse events prior to week 138, 190 and 242
Suspected unexpected serious adverse reactions in longterm follow-up | 242 weeks
  Suspected unexpected serious adverse reactions prior to week 138, 190 and 242

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, Professor, Principal Investigator — IG/MAAG-DARM-LEVER, UZ Leuven, campus Gasthuisberg, Herestraat 49 3000 Leuven
Locations (28):
- Belgium (24):
  - GZA, Antwerp, Antwerpen
  - UZA, Edegem, Antwerpen
  - Erasmus ziekenhuis, Brussels, Brussels Capital
  - Cliniques Universitaires Saint Luc, Brussels, Brussels Capital
  - UZ Brussel, Jette, Brussels Capital
  - CHwapi, Tournai, Henegouwen
  - ZOL Genk, Genk, Limburg
  - CHC Montlégia, Liège, Liège
  - CHU de Liège, Liège, Liège
  - CHU UCL Namur site Godinne, Yvoir, Namur
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Sint lucas Brugge, Bruges, West-Vlaanderen
  - AZ Damiaan, Ostend, West-Vlaanderen
  - OLV Aalst, Aalst
  - Imeldaziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - AZ Sint-Jan, Bruges
  - AZ Sint Lucas, Ghent
  - Jessa ziekenhuis, Hasselt
  - AZ Sint Maarten, Mechelen
  - AZ Delta, Roeselare
  - Vitaz, Sint-Niklaas
- Italy (4):
  - Humanitas research hospital, Milan, Rozzano MI
  - IRCCS De Bellis Castellana Grotte, Castellana Grotte
  - Careggi University Hospital, Florence
  - IRCCS San Raffael Hospital, Milan

IPD SHARING:
Plan to Share IPD: No